CLINICAL TRIAL: NCT02060422
Title: Mindfulness-based Psychotherapy and Social Support Intervention for Drug-resistant Epilepsy
Brief Title: Mindfulness-based Psychotherapy for Drug-resistant Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Venus Tang, Dr, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VP-2011; CRE-2011.167-T (Other: CUHK)
Record Dates: First submitted 2014-02-10; First posted 2014-02-12 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Epilepsy; Stress
Keywords: Epilepsy; Drug-resistant epilepsy; Seizure; Mindfulness; Stress; Psychotherapy
MeSH Terms: conditions — Epilepsy; Drug Resistant Epilepsy; Seizures | interventions — Self-Help Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Social support group (Placebo Comparator): Social support group is an attention-placebo with the same contact hours (four bi-weekly two-and-a-half-hour) as the experimental group, but without active treatment input. The aim of the social support group is to provide a supportive group atmosphere for patients with drug-resistant epilepsy.
  Interventions: Behavioral: Social support group
- Mindfulness-based therapy (Experimental): Mindfulness-based therapy is a four biweekly two-and-a-half-hour psychotherapy tailored for patients with drug-resistant epilepsy. The aims of this therapy are to introduce and practice mindfulness-based stress reduction techniques in coping with drug-resistant epilepsy.
  Interventions: Behavioral: Mindfulness-based therapy

INTERVENTIONS:
Behavioral: Mindfulness-based therapy — Mindfulness-based therapy is a four biweekly two-and-a-half-hour psychotherapy tailored for patients with drug-resistant epilepsy. The aims of this therapy are to introduce and practice mindfulness-based stress reduction techniques in coping with drug-resistant epilepsy.
  Arms: Mindfulness-based therapy
Behavioral: Social support group — Social support group is an attention-placebo with the same contact hours (four bi-weekly two-and-a-half-hour) as the experimental group, but without active treatment input. The aim of the social support group is to provide a supportive group atmosphere for patients with drug-resistant epilepsy.
  Arms: Social support group

SUMMARY:
Psychological problems are prevalent among patients with drug-resistant epilepsy. The bi-directional interaction between psychological well-being and seizure have been recognized in recent years. Reduction of psychological stress has the potential to improve seizure manifestation.

The present study uses an assessor-blinded prospective randomized controlled trial to evaluate the efficacy of a mindfulness-based psychotherapy and an attentional-placebo social support on improving psychological well-being, seizure control and cognitive performance among adult patients with drug-resistant epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of epilepsy
* over 18 years of age
* resistant to pharmacological treatment according to the ILAE guideline
* no previous history of neurosurgery
* adequate level of reading and understanding ability to fill in questionnaires
* capable to communicate with the investigator with considerable expressive capacity
* patients who agree to cooperate with the study procedures required by the protocol
* patients who understand the nature of the study, agree to participate and sign the informed consent form

Exclusion Criteria:

* with primary diagnosis of substance use disorder, mood disorder, bipolar affective disorder, psychosis, or organic mental disorder
* with diagnosis of learning disability or mental retardation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-08; Primary Completion 2013-01 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change in quality of life (Quality of Life in Epilepsy Inventory-31-P Total Score) from baseline to post-intervention | Baseline, 4-week post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Venus Tang, PhD, Principal Investigator — Division of Neurosurgery, Faculty of Medicine, CUHK
Locations (1):
- CUHK Division of Neurosurgery, Faculty of Medicine, Hong Kong, Hong Kong, Hong Kong